CLINICAL TRIAL: NCT03544320
Title: Prediction Using a Randomized Evaluation of Data Collection Integrated Through Connected Technologies for Diabetes Management
Brief Title: Prediction Using Connected Technologies for Diabetes
Acronym: PREDICT-DM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 829150
Record Dates: First submitted 2018-05-18; First posted 2018-06-01 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Pre-Diabetes
Keywords: Pre-diabetes; diabetes; wearable devices; mobile health
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two wearable devices and will wear that device for the duration of the study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The participants will be aware of the two different study arms and the wearable devices used in both. The study investigator will not have not have knowledge of the participants assigned to each arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Activity Monitoring-Wrist worn wearable (Active Comparator): Participants in the activity monitoring-wrist worn wearable group will be randomly assigned to track their activity using a Fitbit Charge 2 for 6 months.
  Interventions: Device: Activity Monitoring-Wrist worn wearable
- Activity Monitoring-Waist-worn wearable (Active Comparator): Participants in the activity monitoring-waist worn wearable group will be randomly assigned to track their activity using a Fitbit Zip for 6 months.
  Interventions: Device: Activity Monitoring-Waist-worn wearable

INTERVENTIONS:
Device: Activity Monitoring-Wrist worn wearable — Participants wear an activity monitor on their wrist.
  Arms: Activity Monitoring-Wrist worn wearable
Device: Activity Monitoring-Waist-worn wearable — Participants wear an activity monitor on their waist.
  Arms: Activity Monitoring-Waist-worn wearable

SUMMARY:
In this study, adults with pre-diabetes will be prospectively enrolled for data collection to design prediction models that integrate electronic health record data and patient-generated activity data. Patients will be randomized to receive either a waist-worn or wrist-worn wearable device for 6 months to capture patient-generated activity data.

DETAILED DESCRIPTION:
Patients with suboptimal glycemic control could be better managed if these higher risk patients could be identified and effective interventions were then targeted towards them. However, most practice settings perform infrequent laboratory testing every 3 to 6 months, if not at longer intervals. Current models to predict change in glycemic control perform poorly and do not take into account the behaviors that occur between these intervals. In this study, we will compare different methods to use data on daily health behaviors collected by wearable devices to enhance risk prediction models. Adults with pre-diabetes will complete a series of surveys and baseline assessments and then will be randomly assigned to use a waist-worn or wrist-worn wearable device for 6 months. Measures of HbA1c and LDL will be obtained at baseline and at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years or older
2. Be able to provide informed consent
3. Have a smartphone or tablet compatible with the wearable device smartphone application and be willing to use the wearable device for 6 months
4. Baseline hemoglobin A1c of 5.7 to 6.4

Exclusion Criteria:

Participants will no be eligible if they have any medical condition or other reason that will likely prohibit them from completing the 6-month study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin A1c | 6 months
  Change in hemoglobin A1c from baseline to 6 months

SECONDARY OUTCOMES:
Change in low-density lipoprotein (LDL) levels | 6 months
  Change in LDL level from baseline to 6 months

OTHER OUTCOMES:
Hospitalization | 6 months
  Admission to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh S Patel, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Medicine, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No